CLINICAL TRIAL: NCT05380115
Title: Implementation of Cognitive-behavioral Therapy for Older Adults With Generalized Anxiety Disorder
Brief Title: Cognitive Behavioral Therapy (CBT) for Late Life Anxiety
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators were running out of time on a 1 year pilot grant and had to prioritize other parts of the study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00084483
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: late-life anxiety; aging; cognitive-behavioral therapy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT (Experimental): All subjects enrolled received CBT for 10 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — weekly one on one video or telephone interviews with a study coach

SUMMARY:
The purpose of this research study is to assess the acceptability and feasibility of the implementation strategy and fidelity of cognitive-behavioral therapy (CBT) for older adults with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
All participants will receive CBT. Each subject will be given a workbook and each chapter in the workbook provides information about a different coping strategy for managing worry and anxiety. There will be a daily assignment in the workbook to complete before a call with the personal study coach. For 10 weeks, participants will have a 45-50 minute session (telephone or video) each week with their study coach. These calls will be confidential. The participant and the personal study coach will review the assigned chapter and completed homework during the weekly telephone sessions. Participants will also fill out questionnaires before starting sessions, when completing all 10 sessions, and 6 months after completing sessions.

ELIGIBILITY:
Inclusion Criteria:

* participants who have had an outpatient visit to an Atrium provider
* at least one of the following: any diagnosis of an anxiety or depressive disorder; anxiety, depression, or sleep disturbance as a symptom in the problem list or in the note; and use of anxiolytic, anti-depressant, and sleep aide medications.

Exclusion Criteria:

* diagnosis of dementia or cognitive impairment in the problem list

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder scale (GAD-7) | Week 11
  Self-report measure of GAD symptoms. Total scores can range from 0 to 21; higher scores indicate more GAD symptoms.
Penn State Worry Questionnaire-Abbreviated (PSWQ-A) | week 11
  8-item measure of frequency/intensity of worry; most commonly used worry measure. Scores can range from 8 to 40; higher scores indicate higher levels of worry.
Feasibility-Expectancy Rating Scale | Week 1
  Assesses beliefs in how logical the treatment received seems, confidence in undergoing treatment/recommending to others, and expectations for success. Used in anxiety treatment studies with older adults. Scores can range from 4 to 40; higher scores indicate more positive expectations.
Feasibility-Intervention adherence | Week 11
  The percentage of completed sessions
Feasibility-Number of participants who complete at least 75% of sessions | Week 11

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | baseline, week 6, week 11
  8-item measure of general anxiety symptoms; each item is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always); scores can range from 8 to 40; higher scores indicate greater severity of anxiety.
Insomnia Sleep Index | baseline, week 6, week 11
  7-item self-report measure of type and severity of insomnia symptoms. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem); scores can range from 0 to 28 with higher scores indicating more severe insomnia.
Feasibility-Client Satisfaction Questionnaire | Week 11
  Assesses satisfaction with treatment. Scores can range from 8 to 32; higher scores indicate more satisfaction.
Feasibility-Working Alliance Inventory, Client | Week 11
  Assesses therapist-client working alliance. 12 items on a 7-point scale (1=never; 7=always); scores can range from 12 to 84 with higher scores indicating better working relationship.
Feasibility-Working Alliance Inventory, Therapist | Week 11
  Assesses therapist-client working alliance. 12 items on a 7-point scale (1=never; 7=always); scores can range from 12 to 84 with higher scores indicating better working relationship.
Generalized Anxiety Disorder scale (GAD-7) | Baseline
  Self-report measure of GAD symptoms. Total scores can range from 0 to 21; higher scores indicate more GAD symptoms.
Generalized Anxiety Disorder scale (GAD-7) | Week 6
  Self-report measure of GAD symptoms. Total scores can range from 0 to 21; higher scores indicate more GAD symptoms.
Penn State Worry Questionnaire-Abbreviated (PSWQ-A) | baseline
  8-item measure of frequency/intensity of worry; most commonly used worry measure. Scores can range from 8 to 40; higher scores indicate higher levels of worry.
Penn State Worry Questionnaire-Abbreviated (PSWQ-A) | week 6
  8-item measure of frequency/intensity of worry; most commonly used worry measure. Scores can range from 8 to 40; higher scores indicate higher levels of worry.

OTHER OUTCOMES:
Healthcare Utilization-Number of Outpatient encounters | Week 37
Healthcare Utilization-Number of ED visits | Week 37
Healthcare Utilization-Number of inpatient stays | Week 37
Healthcare Utilization-Costs for outpatient encounters, ED visits and inpatient stays | Week 37
Qualitative Interviews | Week 11
  Analyses will be primarily conducted by Q-PRO

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Brenes, PhD, Principal Investigator — Atrium Health Wake Forest Baptist

IPD SHARING:
Plan to Share IPD: No